CLINICAL TRIAL: NCT04889404
Title: LYNPARZA Tablets 100 mg, 150mg General Drug Use-results Study in Patients on Maintenance Treatment After Platinum-based Chemotherapy for BRCA Mutated Curatively Unresectable Pancreas Cancer
Brief Title: LYNPARZA Pancreas Cancer Japan Post-Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D081FC00004
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To collect and characterise the incidence of adverse events related to the safety specifications of the maintenance treatment after platinum-based chemotherapy in patients with BRCA mutated pancreatic cancer under the actual post-marketing use of LYNPAZA.

DETAILED DESCRIPTION:
To collect and characterise the incidence of adverse events related to the safety specifications*1 of the maintenance treatment after platinum-based chemotherapy in patients with BRCA mutated pancreatic cancer under the actual post-marketing use of LYNPAZA.

This investigation will be conducted for application for re-examination specified in Article 14-4 of the Pharmaceutical Affairs Law.

*1: Bone marrow depression, interstitial lung disease, new primary malignancies, and embryofoetal toxicity

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive LYNPARZA for the first time for the maintenance treatment after platinum-based chemotherapy in patients with BRCA mutated curatively unresectable pancreas cancer after the approval date of partial change application for the additional indication (25/Dec./2020).

Exclusion Criteria:

* Patients who have no treatment history with LYNPARZA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients on maintenance treatment after platinum-based chemotherapy for BRCA mutated curatively unresectable pancreas cancer
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to the safety specifications | from baseline to 1year
  Safety specifications:Bone marrow depression, interstitial lung disease, new primary malignancies, and embryofoetal toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — Astrazeneca KK
Locations (60):
- Japan (60):
  - Research Site, Osaka, Lyn010001
  - Research Site, Kanagawa, Lyn010003
  - Research Site, Okayama, Lyn010004
  - Research Site, Akita, Lyn010005
  - Research Site, Niigata, Lyn010006
  - Research Site, Shizuoka, Lyn010007
  - Research Site, Niigata, Lyn010008
  - Research Site, Tokyo, Lyn010009
  - Research Site, Saitama, Lyn010010
  - Research Site, Aichi, Lyn010011
  - Research Site, Osaka, Lyn010012
  - Research Site, Tokyo, Lyn010013
  - Research Site, Nara, Lyn010014
  - Research Site, Wakayama, Lyn010015
  - Research Site, Miyagi, Lyn010016
  - Research Site, Tokyo, Lyn010017
  - Research Site, Osaka, Lyn010018
  - Research Site, Gunma, Lyn010019
  - Research Site, Hiroshima, Lyn010020
  - Research Site, Tochigi, Lyn010021
  - Research Site, Numakunai, Lyn010022
  - Research Site, Osaka, Lyn010025
  - Research Site, Shizuoka, Lyn010026
  - Research Site, Nagasaki, Lyn010027
  - Research Site, Kumamoto, Lyn010028
  - Research Site, Saitama, Lyn010029
  - Research Site, Nagano, Lyn010031
  - Research Site, Hyōgo, Lyn010032
  - Research Site, Shimane, Lyn010033
  - Research Site, Hyōgo, Lyn010034
  - Research Site, Shizuoka, Lyn010035
  - Research Site, Hyōgo, Lyn010036
  - Research Site, Okayama, Lyn010038
  - Research Site, Fukuoka, Lyn010041
  - Research Site, Hokkaido, Lyn010042
  - Research Site, Ehime, Lyn010044
  - Research Site, Osaka, Lyn010045
  - Research Site, Shizuoka, Lyn010047
  - Research Site, Tokyo, Lyn010050
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kyoto
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Shizuoka
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081FC00004&attachmentIdentifier=dc30d268-3cc6-453e-880a-c614385118e4&fileName=Lynparza_Japan_PARCS_D081FC00004_CSR_Synopsis.pdf&versionIdentifier=